CLINICAL TRIAL: NCT00790764
Title: Phase II Study for the Transfer of Bone Marrow-Derived Mononuclear and Mesenchymal StemCells Into the Myocardium for the Treatment of Severe Coronary Ischemia
Brief Title: Phase II Combination Stem Cell Therapy for the Treatment of Severe Coronary Ischemia(CI)
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Suspended due to lack of funding.
Sponsor: TCA Cellular Therapy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008--03-II
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2011-04

CONDITIONS: Heart Disease; Blocked Arteries; Coronary Ischemia; Coronary Disease; Coronary Artery Disease; Coronary Atherosclerosis
MeSH Terms: conditions — Heart Diseases; Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 20 individuals will receive placebo.
  Interventions: Other: placebo
- MESENDO (Experimental): Active combination autologous stem cell therapy. 40 individuals will receive MESENDO in either the "high" or "low" dose treatment groups.
  Interventions: Biological: MESENDO

INTERVENTIONS:
Biological: MESENDO — For the cell product, proper aliquots of each cell type will be taken to fulfill the doses established for this protocol. The two aliquots will be mixed and resuspended to a final volume of 3 ml in the 'Final Suspension Medium' which consists of Dulbecco's Phosphate Buffered Saline (DPBS), containing 5% human serum albumin.
  Arms: MESENDO
Other: placebo — For placebo, 3 ml of the 'Final Suspension Medium' which consists of Dulbecco's Phosphate Buffered Saline (DPBS), containing 5% human serum albumin will be transferred to a 5 ml syringe
  Arms: Placebo

SUMMARY:
The present investigation will be a Phase II, single center, placebo-controlled, randomized, dose escalation, infusion modality (intracoronary vs transendocardial injection using the Cordis Biosense NOGASTAR TM Mapping Catheter with the Biosense MYOSTAR TM left ventricular injection catheter) transplantation of an autologous (your own stem cells) combination of bone marrow-derived stem cells into myocardium for the treatment of severe coronary ischemia.

The purpose of this research study is to determine if the infusion of a combination of stem cells obtained from the bone marrow of the same patient will contribute to the formation of new blood vessels in patients with symptomatic severe coronary ischemia(CI).

In this trial we will determine whether the combination stem cell treatment is safe, feasible and results in the development of mature stable and/or collateral vessels and improvement of cardiac function.

Coronary Ischemia (CI) is intractable angina due to severe coronary artery disease which can seriously decrease blood flow to the heart.

CI needs a comprehensive treatment since the condition will not improve on its own. The overall goal of the treatment is to increase blood flow to the heart and improve symptoms of angina.

The study hypothesis is based on the concept that the process of formation of new blood vessels is complex and requires the participation of several types of stem cells and growth factors. The lack of any of these components will produce vessels which are immature and unable to provide appropriate blood supply to the heart.

Patients eligible to participate in this study are those suffering from severe blockages of the vessels of the heart and are not candidates for percutaneous revascularization or surgical procedures.

DETAILED DESCRIPTION:
Enrolled individuals (60) will be divided in 2 Treatment groups for the infusion of the cell /placebo product:

1. Treatment Group A (30 individuals, including patients and placebo controls) will receive the product by intracoronary infusion,
2. Treatment Group B (30 individuals, including patients and placebo controls) will receive the product by transendocardial injections.

   In turn, each Treatment Group will consist of 2 subgroups of individuals that will receive the infusion of one of the two doses established of the cell product:
3. In treatment SubGroup 1, 10 individuals will receive the "low dose" of the cell product and 5 individuals will receive the placebo product.
4. In treatment SubGroup 2, 10 individuals will receive the "high dose" of the cell product and 5 individuals will receive the placebo product

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80
* Male or female
* Angina pectoris: Canadian Cardiovascular Society Class III or IV or symptoms consistent with angina equivalent (dyspnea) CCS Class III or IV (Functional Class)
* Chronic coronary artery disease in at least one epicardial vessel with stenosis > 70% by coronary angiography within the last 6 months
* Stable medical therapy for at least one month
* Reversible perfusion defects by SPECT
* Not a candidate for coronary artery by-pass surgery due to poor targets or small vessels and not a candidate for percutaneous intervention due to small vessels or unreachable coronary lesions due to complicated anatomy

Exclusion Criteria:

* Inability to give written informed consent
* Previous angiogenic therapy or myocardial laser therapy
* Recent (< 4 weeks) acute ST-elevation myocardial infarction
* Patients with severe valvular heart disease
* Recent malignancy or radiation therapy (< 6 months) and not expected to survive 6 months
* Known sensitivity to gentamycin and/or amphotericin B
* Use or expected use of antineoplastic drugs
* Renal insufficiency with creatinine greater than 2.7 unless on dialysis
* WBC greater than 13,000 or lower than 3,000
* Hematocrit lower than 30 or higher than 50
* Platelet counts lower than 60,000 or higher than 500,000
* Child bearing potential without use of contraceptives
* Pregnant or planning to become pregnant
* Any illness which, in the investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient's safety, or interfere with the interpretation of the sturdy results
* Any illness which might affect patient's survival over the study follow-up period
* History of skeletal muscle disease, either primary (i.e. myopathy) or secondary (i.e. ischemic) or any underlying myopathy such as myasthenia gravis, muscular dystrophy, etc
* Patients with active infectious disease and/or who are known to have tested positive for HIV, HTLV, HBV-sAg, HCV, AST or ALT > 2 times ULRR
* Cardiogenic shock
* Any significant laboratory abnormality which will in the investigator's opinion interfere with the patient's ability to comply with the protocol, compromise the patient's safety, or interfere with the interpretation of the study result

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-11; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by laboratory assessments, ecg and temperature. | 2 weeks

SECONDARY OUTCOMES:
Efficacy as measured by SPECT scan, MUGA scan and 2D Echogradiogram | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel P. Lasala, MD, Principal Investigator — TCA Cellular Therapy
Locations (1):
- TCA Cellular Therapy, Covington, Louisiana, United States